CLINICAL TRIAL: NCT01385852
Title: Impact of Different Fluidic Parameters on Development of Cystoid Macular Edema Following Phacoemulsification
Brief Title: CME With Different Fluidic Parameters
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Iladevi Cataract and IOL Research Center (Other)
Responsible Party: Principal Investigator, Abhay R. Vasavada, principal investigator, Iladevi Cataract and IOL Research Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 10-005
Record Dates: First submitted 2011-06-28; First posted 2011-06-30 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-06

CONDITIONS: Cystoid Macular Edema Following Cataract Surgery
Keywords: CME; OCT; Optical coherence tomography; macular thickness
MeSH Terms: interventions — Phacoemulsification

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Longitudinal U/S - low fluidic (Active Comparator): ASPIRATION FLOW RATE - 25 CC/MIN, BOTTLE HEIGHT - 90 CMS, LONGITUDINAL ULTRASOUND
  Interventions: Procedure: microcoaxial phacoemulsification
- Torsional U/S - low fluidic (Active Comparator): ASPIRATION FLOW RATE - 25 CC/MIN, BOTTLE HEIGHT - 90 CMS, TORSIONAL ULTRASOUND
  Interventions: Procedure: microcoaxial phacoemulsification
- Longitudinal U/S - high fluidic (Active Comparator): ASPIRATION FLOW RATE - 40 CC/MIN, BOTTLE HEIGHT - 110 CMS, LONGITUDINAL ULTRASOUND
  Interventions: Procedure: microcoaxial phacoemulsification

INTERVENTIONS:
Procedure: microcoaxial phacoemulsification — conventional longitudinal ultrasound
  Other Names: phacoemulsification; small incision cataract surgery

SUMMARY:
Understanding and modulating fluid parameters is an important, but often overlooked aspect of phacoemulsification. In a previous study we compared the impact of using high fluid parameters versus low fluidic parameters on real-time IOP measured during phacoemulsification. The investigators found that using high parameters resulted in a higher absolute rise in IOP as well as higher fluctuations in the IOP when compared to low parameters. Clinically these higher fluctuations in IOP would translate in a higher chamber instability. Based on the results of this study, the investigators decided to take it further and study the impact of using high parameters (and thus, higher chamber instability) on macular edema and thickness following surgery, in an otherwise uncomplicated surgery.

Higher fluid parameters during phacoemulsification predisposes the eye to increased macular thickness

DETAILED DESCRIPTION:
Several studies have shown the adverse impact of an increase in the IOP and IOP fluctuations that occur during anterior segment intervention on the posterior segment structures. In human volunteers with each incremental increase in IOP the systolic and diastolic flow velocities in the short posterior ciliary arteries decreased linearly. This implies that the normal healthy eye is not able to autoregulate to maintain posterior ciliary artery blood flow velocities in response to acute large elevations in IOP. Vascular insufficiency due to abnormal autoregulation has been proposed as a major factor in the development of glaucoma. 1

It has been postulated that IOP elevation during the LASIK procedure causes mechanical stress which may induce tangential stress on the posterior segment.2, 3 Some studies have reported that the increase in IOP damages the retinal ganglion cells causing visual field defects. Also sudden increases in IOP, although well tolerated may induce changes in the peripheral retina.4,5,6

Several reports propose the occurrence of macular hole, lacquer cracks and choroidal neovascular membranes following the LASIK procedure. 3 It has been observed that the rapidly fluctuating pressure variations may be detrimental, particularly in susceptible persons with compromised ocular blood flow. Rapid IOP changes across a 30-mm Hg range would be predicted to influence posterior segment blood vessels.

In a previous study we compared the impact of using high fluid parameters versus low fluidic parameters on real-time IOP measured during phacoemulsification. We found that using high parameters resulted in a higher absolute rise in IOP as well as higher fluctuations in the IOP when compared to low parameters. Clinically these higher fluctuations in IOP would translate in a higher chamber instability.

We hypothesize that although transient, the increased IOP that occurs during phacoemulsification when using high parameters could cause mechanical stress on the eye. These higher fluid parameters during phacoemulsification can predispose the eye to increased macular thickness.

To the best of our knowledge there are no published data on impact of IOP changes and fluctuation that are induced during cataract surgery on the macula. To investigate this further, we decided to study the impact of using high parameters (and thus, higher chamber instability) on macular thickness following surgery, in an otherwise uncomplicated surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Uncomplicated, Age-related cataract.
2. Nuclear sclerosis: upto grade 3
3. Age: 40-70 years
4. Axial length: 21.5 mm to 24.5 mm

Exclusion Criteria:

1. Diabetes mellitus
2. Co-existing ocular disease- uveitis, glaucoma, PEX
3. Pre-existing macular pathology (eg.ARMD)
4. Previously operated eyes
5. Under treatment with Topical or systemic steroids / NSAID's
6. Intraoperative complications- PCR, Descemet's detachment, uveal trauma
7. Post operative complications - severe inflammation (>grade 3), rise in IOP

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2010-05; Primary Completion 2011-02 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
cystoid macular edema (CME) | 3 months
  A > or = 30% increase in baseline central foveal thickness measaured by anterior segment OCT will be defined as having CME.

SECONDARY OUTCOMES:
macular thickness | 1, 3 months
  macular thickness measured in 3 zones using the anterior segment OCT
central corneal thickness (CCT) | first post-operative day,
  CCT will be measured on the ultrasound pachymeter by a single experienced observer
endothelial cell loss | 6 months post-operative
  Endothelial cell loss will be measured using a specular microscope in the central area by a single technician
anterior chamber inflammation | 1 months
  it will be assessed on the slit lamp examination by a single experienced observer using the Hogan's criteria
CORRECTED DISTANCE VISUAL ACUITY (CDVA) | 3 months
  visual acuity (VA) of 20/40 or worse was defined as "clinically significant"

CONTACTS AND LOCATIONS:
Overall Officials: ABHAY R VASAVADA, MS, FRCS, Principal Investigator — ILADEVI CATARACT AND RESEARCH CENTER
Locations (1):
- Raghudeep Eye Clinic, Ahmedabad, Gujarat, India

REFERENCES:
- [Result] Kim SJ, Belair ML, Bressler NM, Dunn JP, Thorne JE, Kedhar SR, Jabs DA. A method of reporting macular edema after cataract surgery using optical coherence tomography. Retina. 2008 Jun;28(6):870-6. doi: 10.1097/IAE.0b013e318169d04e. PMID 18536605
- [Result] Cagini C, Fiore T, Iaccheri B, Piccinelli F, Ricci MA, Fruttini D. Macular thickness measured by optical coherence tomography in a healthy population before and after uncomplicated cataract phacoemulsification surgery. Curr Eye Res. 2009 Dec;34(12):1036-41. doi: 10.3109/02713680903288937. PMID 19958122
- [Result] Belair ML, Kim SJ, Thorne JE, Dunn JP, Kedhar SR, Brown DM, Jabs DA. Incidence of cystoid macular edema after cataract surgery in patients with and without uveitis using optical coherence tomography. Am J Ophthalmol. 2009 Jul;148(1):128-35.e2. doi: 10.1016/j.ajo.2009.02.029. Epub 2009 Apr 29. PMID 19403110
- [Result] Lee YC, Chung FL, Chen CC. Intraocular pressure and foveal thickness after phacoemulsification. Am J Ophthalmol. 2007 Aug;144(2):203-208. doi: 10.1016/j.ajo.2007.04.020. Epub 2007 May 30. PMID 17540324
- [Result] Kim SJ, Equi R, Bressler NM. Analysis of macular edema after cataract surgery in patients with diabetes using optical coherence tomography. Ophthalmology. 2007 May;114(5):881-9. doi: 10.1016/j.ophtha.2006.08.053. Epub 2007 Feb 1. PMID 17275910
- [Result] Perente I, Utine CA, Ozturker C, Cakir M, Kaya V, Eren H, Kapran Z, Yilmaz OF. Evaluation of macular changes after uncomplicated phacoemulsification surgery by optical coherence tomography. Curr Eye Res. 2007 Mar;32(3):241-7. doi: 10.1080/02713680601160610. PMID 17453944
- [Result] Biro Z, Balla Z, Kovacs B. Change of foveal and perifoveal thickness measured by OCT after phacoemulsification and IOL implantation. Eye (Lond). 2008 Jan;22(1):8-12. doi: 10.1038/sj.eye.6702460. Epub 2006 Jun 2. PMID 16751754